CLINICAL TRIAL: NCT06304597
Title: Improving Detection and Treatment of Locally Advanced Rectal Cancer by Dual Wavelength Quantitative Fluorescence Molecular Endoscopy Using Nivolumab-800CW and Durvalumab-680LT
Brief Title: Evaluating PD-1/PD-L1 in Locally Advanced Rectal Cancer by Quantitative Fluorescence Molecular Endoscopy
Acronym: PREDICT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17651
Record Dates: First submitted 2023-11-14; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced Rectal Carcinoma
MeSH Terms: interventions — durvalumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab-680LT and nivolumab-800CW (Experimental): Study procedure 1: Combined intravenous tracer administration with 15mg IMFINZI and 15mg OPDIVO followed by fluorescence molecular endoscopy
  Study procedure 2: Combined intravenous tracer administration with 15mg IMFINZI and 15mg OPDIVO followed by fluorescence molecular endoscopy
  Interventions: Drug: Imfinzi; Drug: Opdivo

INTERVENTIONS:
Drug: Imfinzi — Durvalumab is labeled to IRDye-680LT and will be administered in combination with fluorescently labelled nivolumab (Opdivo)
  Other Names: durvalumab
Drug: Opdivo — Nivolumab is labeled to IRDye-800CW and will be administered in combination with fluorescently labelled durvalumab (Imfinzi)
  Other Names: Nivolumab

SUMMARY:
Colorectal cancer (CRC) claims 10% of global cancer-related deaths annually, with rising incidence. Locally advanced rectal cancer (LARC) requires improved diagnostic techniques. This study focuses on dual-wavelength quantitative fluorescence molecular endoscopy (qFME) using PD-1/PD-L1-targeted tracers for LARC patients undergoing neoadjuvant treatment. Eighteen patients will receive nivolumab-800CW and durvalumab-680LT before qFME procedures, assessing programmed death-1/programmed death ligand-1 (PD-1/PD-L1) expression. We want to test the feasibility of qFME and ex vivo fluorescence imaging after intravenous administration of nivolumab-800CW, targeting PD-1, and durvalumab-680LT, targeting PD-L1, to visualize PD-L1 and PD-1 expression before and after CRT in LARC patients. If successful, this method can potentially be used in the future to see which patients most likely benefit from additional immunotherapy beforehand. The non-randomized, prospective phase 1 intervention explores biomarkers' role in treatment response prediction. Tracer administration poses minimal risks. Patients will not directly benefit, but the study aims to establish the utility of nivolumab-800CW and durvalumab-680LT in determining PD-1/PD-L1 expression during endoscopy.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) constitutes a significant global health burden, responsible for 10% of cancer-related deaths annually, with incidence rates escalating by 1-4% annually. Locally advanced rectal cancer (LARC) demands enhanced diagnostic tools, despite various existing modalities. This prospective, non-randomized, phase 1 intervention study addresses this need through dual-wavelength quantitative fluorescence molecular endoscopy (qFME) utilizing PD-1/PD-L1-targeted tracers. The primary goal is to assess the safety and feasibility of using durvalumab-680LT and nivolumab-800CW to assess PD-1 and PD-L1 expression alterations before and after neoadjuvant chemoradiotherapy (nCRT) in LARC patients.

The study's central hypothesis posits that higher PD-1/PD-L1 expression correlates with improved treatment response. To test this, eighteen LARC patients scheduled for nCRT and surgery will receive intravenous nivolumab-800CW and durvalumab-680LT, with qFME procedures conducted before and after nCRT. The tracers, labeled with different near-infrared (NIR) fluorophores (800CW and 680LT), allow separate quantification during simultaneous administration.

The study design is single-center, non-blinded, and non-randomized. Eligible patients, identified at the University Medical Center Groningen (UMCG), undergo qFME during staging endoscopy pre-nCRT and an additional procedure 2-3 weeks post-nCRT. Tracer administration precedes these procedures, involving monitoring for potential side effects. A potential third restaging endoscopy occurs 6-8 weeks post-CRT, without tracer administration, collecting biopsies.

The study population comprises eighteen LARC patients (cT3c-4, N1-2, M0) at UMCG scheduled for nCRT followed by surgery. Tracer administration involves 15 mg nivolumab-800CW and 15 mg durvalumab-680LT, with endoscopy procedures incorporating high-definition white-light endoscopy (HD-WLE), qFME, multi-diameter single fiber reflectance/single fiber fluorescence (MDSFR/SFF) spectroscopy, endoscopic rectal ultrasound (EUS), fine needle aspiration (FNA) biopsy, and ultrasound-guided needle biopsy single-fiber fluorescence (USNB/SFF) spectroscopy.

The main study parameters assess the safety of the combination of durvalumab-680LT and nivolumab-800CW through the evaluation of both vital signs after tracer administration and possible (severe) adverse events (SAE/AE's). Importantly, we will determine the feasibility of fluorescence molecular imaging using the GMP-produced near-infrared fluorescent tracers durvalumab-680LT and nivolumab-800CW for visualizing PD-1 and PD-L1 expression before and after nCRT in LARC patients with dedicated fluorescence imaging systems. Risks include minimal infection and hematoma risks from tracer administration, and the study offers negligible benefits to participants. The study's significance lies in establishing the utility of nivolumab-800CW and durvalumab-680LT in determining PD-1/PD-L1 expression during endoscopy for potential treatment response prediction in LARC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with LARC (cT3c-4, N1-2, M0);
* Written informed consent is obtained; (We aim to include only patients who consent to both study procedures, however if some patients (n<9) do not consent to the first or second procedure or withdraw their consent for the second procedure after the first procedure, they can still be included)
* Be at least 18 years old;
* Speak the Dutch language.

Exclusion Criteria:

* Concurrent uncontrolled medical conditions according to treating medical physician;
* Pregnancy or breast feeding. A negative pregnancy test must be available for women of childbearing potential on the day of tracer administration (i.e. premenopausal women with intact reproductive organs and women less than two years after menopause);
* Prior irradical endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) of the primary tumor.
* Received an investigational drug within 30 days prior to administration of nivolumab-800CW and durvalumab-680LT according to the patient's medical history;
* History of infusion reactions to nivolumab, durvalumab or other monoclonal antibodies according to the patient's medical history;
* Active episode of inflammatory bowel disease;
* Use of immunosuppressive agents;
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent according to treating medical physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety of nivolumab-800CW in combination with durvalumab-680LT | Until 24 hours after administration
  To evaluate the safety of nivolumab-800CW in combination with durvalumab-680LT through monitoring vital signs, the injection site and evaluating possible tracer-related (severe) adverse events (SAE/AEs) and suspected unexpected serious adverse reactions (SUSARs).
To investigate the feasibility of using fluorescence molecular endoscopy (FME) and ex vivo FMI to detect nivolumab-800CW and durvalumab-680LT signals indicating PD1 and PD-L1 expression. | 12 months
  Determine in vivo fluorescent signal in tumor and surrounding tissue by noting yes/no and the number of lesions detected by HD-WLE and qFME on recorded location during the endoscopic procedure. Semi-quantification of signal intensities of different areas by collecting the mean and standard deviation for the targeted area and surrounding tissue (looking at intra and inter variability). Afterwards comparisons of TBRs/CNRs can be performed. Durvalumab-680LT and nivolumab-800CW detection by fluorescence microscopy (yes/no). Mean fluorescence intensity (MFI) calculation of biopsies Quantified PD-L1/PD-1 expression by qPCR and Western Blot will be correlated to in vivo fluorescence signals, MDSFR/SFF measurements and MFI calculations of biopsies.
Heart rate | Until 24 hours after administration
  Beats per minute
Blood pressure systolic and diastolic | Until 24 hours after administration
  Millimeters of mercury (mmHg)
Temperature | Until 24 hours after administration
  Degrees Celsius

SECONDARY OUTCOMES:
Determine the PD-1 and PD-L1 expression and the changes in PD-1 and PD-L1 expression before and after nCRT in patients with LARC. | 12 months
  Quantified PD-L1/PD-1 expression by qPCR will be compared before and after CRT.
Determine the PD-1 and PD-L1 expression and the changes in PD-1 and PD-L1 expression before and after nCRT in patients with LARC. | 12 months
  Quantified PD-L1/PD-1 expression by Western Blot will be compared before and after CRT.
Quantify in vivo fluorescence signals of nivolumab-800CW and durvalumab-680LT before and after CRT by using MDSFR/SFF spectroscopy/UNSB/SFF spectroscopy and correlate these measurements to, in vivo fluorescence intensities and PD1/PD-L1 expression | 12 months
  Evaluation of staining intensities by scored positive/negative in percentages and the H-score will be calculated by two independent researchers to evaluate staining intensities. qPCR and Western Blot quantifications (numerical values) will be compared to H-scores.
Quantify in vivo fluorescence signals of nivolumab-800CW and durvalumab-680LT before and after CRT by using MDSFR/SFF spectroscopy/UNSB/SFF spectroscopy and correlate these measurements to, in vivo fluorescence intensities and PD1/PD-L1 expression | 12 months
  qPCR and Western Blot quantifications and H-scores will be correlated to MDSFR/SFF spectroscopy/UNSB/SFF spectroscopy measurements
Perform real-time polymerase chain reaction (qPCR) and western blot on biopsies to determine whether there is genetic downregulation or protein degradation of PD-1 and PD-L1 after chemoradiotherapy | 12 months
  qPCR and Western Blot quantifications (numerical values) will be compared to each other
Compare immune cell composition between the radiated and non-radiated area of the bowel. | 12 months
  Immune cell composition (percentages)measured by FACS will be compared in biopsies from radiated and non radiated areas and in the blood from before and after CRT.
Evaluate targeted detection with nivolumab-800CW and durvalumab-680LT of the tumor by ex vivo visualization of the resection specimen with PEARL Trilogy | 12 months
  Fluorescence of the resection specimen will be measured with the PEARL Trilogy

CONTACTS AND LOCATIONS:
Overall Officials: Wouter B Nagengast, Prof., Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No